CLINICAL TRIAL: NCT07281807
Title: Comparison of the Pain Levels of Single-Dose Premedication With Piroxicam and Prednisolone on Post-Endodontic Pain in Single-Visit Root Canal Treatment of Premolars
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RANA AHMAD (Other)
Responsible Party: Sponsor-Investigator, RANA AHMAD, Dr, Shaheed Zulfiqar Ali Bhutto Medical University
Organization: Shaheed Zulfiqar Ali Bhutto Medical University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TUF/IRB/28/2025
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Irreversible Pulpitis With Apical Periodontitis; Symptomatic Apical Periodontitis
MeSH Terms: interventions — Premedication; Piroxicam

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A: piroxicam (Experimental): Group A: patients will be given piroxicam 20mg as premedication
  Interventions: Drug: piroxicam 20mg
- Group B: prednisolone (Active Comparator): Group B: patients will be given prednisolone 20mg as premedication
  Interventions: Drug: Group B: patients will be given prednisolone 20mg as premedication

INTERVENTIONS:
Drug: Group B: patients will be given prednisolone 20mg as premedication — Group B: patients will be given prednisolone 20mg as premedication
  Arms: Group B: prednisolone
Drug: piroxicam 20mg — Group A: patients will be given piroxicam 20mg as premedication
  Arms: Group A: piroxicam

SUMMARY:
To compare the post operative mean pain scores by administering single-dose preoperative piroxicam and prednisolone in patients of irreversible pulpitis with symptomatic apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patient ranging between 18-40 years
* Having at least one premolar with diagnosis of symptomatic irreversible pulpitis according to history, examination and radiographs.
* Teeth having mature apex confirmed by periapical radiographs.

Exclusion Criteria:

* History of systemic disorders including HIV, Hepatitis

  * Pregnancy (As per Medical record/ Verbally)
  * Patient using medication such as analgesics or anti-inflammatory drugs
  * Patient allergic to lignocaine, piroxicam and prednisolone
  * Tooth not suitable for restoration
  * Periodontal probing depth ≥ 4mm
  * Retreatment cases
  * Patients having calcified canals assessed by radiographic findings

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
pain after single visit root canal treatment | 48 hours
  pain score on visual analogue scale

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vatankhah M, Zargar N, Naseri M, Salem S, Baghban AA, Etemadi A, Dianat O. Analgesic Efficacy of Ibuprofen and Diclofenac Potassium on Postoperative Endodontic Pain in Maxillary and Mandibular First Molars with Irreversible Pulpitis: A Randomised Controlled Trial. Eur Endod J. 2023 Mar;8(2):133-139. doi: 10.14744/eej.2022.45238. PMID 37010198
- [Result] Benkhalil AM, Rmdan GA. Effect of Prednisolone Premedication on Postoperative Pain after Single Visit Endodontic Therapy: A Randomized Controlled Trial. Sch J App Med Sci. 2022;8:1219-26.